CLINICAL TRIAL: NCT03160313
Title: Effects of an Interdisciplinary Fitness and Social Engagement Intervention on Physical Activity, Sleep Quality and Community Integration
Brief Title: Effects of an Interdisciplinary Fitness and Social Engagement Intervention
Acronym: InFuSe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01798
Record Dates: First submitted 2017-03-28; First posted 2017-05-19 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Social engagement; Physical Activity; Sleep Quality; Traumatic Brain Injury; Veteran
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InFuSE (Experimental): Experimental group which will receive health education, group discussion, and supervised exercise.
  Interventions: Behavioral: InFuSE
- Patient Education/Group Discussion (Active Comparator): Active control group which will receive health education and group discussion.
  Interventions: Behavioral: Patient Education/Group Discussion

INTERVENTIONS:
Behavioral: InFuSE — Each session includes a 45-minute education and group discussion. A 60-minute exercise component then completes the session. Each topic was specifically picked and tailored to benefit Veterans with TBI. The education sessions will be led and moderated by different professionals including physical therapists, recreation therapists, and physicians. Participants will be asked to participate in several learning activities. The activities are included to help improve understanding and promote group discussion. The exercise piece consists of a warm-up, endurance training (20-30 minutes), strengthening (15 minutes), balance/cognitive training (15 minutes), and a cool-down.
  Arms: InFuSE
Behavioral: Patient Education/Group Discussion — Each week you will participate in a 1 hour health education class with other Veterans. Each topic was specifically picked and tailored for Veterans with TBI. These education sessions will be led and moderated by different professionals including physical therapists, recreation therapists, and physicians. Participants will be asked to participate in several learning activities which are included to help improve understanding and promote group discussion.
  Arms: Patient Education/Group Discussion

SUMMARY:
This study will evaluate feasibility and preliminary effectiveness of a 10-week interdisciplinary and multimodal intervention that utilizes patient education, group discussion, and supervised exercise for Veterans with a history of traumatic brain injury (TBI). Primary outcomes include physical activity (PA), sleep quality, and community integration.

DETAILED DESCRIPTION:
This randomized controlled trial will have a sample size of 24. Veterans between the ages of 18 and 65 in the Polytrauma and TBI program who are greater than 1 year post injury prior to entering the study, will be recruited. After randomization participants in the intervention group will complete a 10 week bout of multidisciplinary wellness education, group discussion, and supervised exercise. The intervention will occur weekly and last up to 2 hours. The control group will complete a 10week comprehensive health education program simultaneously. All measures will be collected again, post intervention. A follow-up collection will occur at 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* TBI of at least mild severity using criteria related to disturbance of consciousness
* Most recent TBI occurred >1 year prior to consent process
* Medically stable with physician approval to participate

Exclusion Criteria:

* Unable to provide informed consent and no proxy available
* Prior history of known bipolar disorder or schizophrenia or severe psychiatric illness
* Veterans with any cardiac condition that may cause sudden decompensation during cardiovascular testing and training (e.g., severe congestive heart failure and uncontrolled hypertension)
* Veteran is currently active in a skilled physical therapy program.
* Veterans who meet or exceed American Heart Association and American College of Sports Medicine guidelines for physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Exercise Self-Efficacy Scale (ESES) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  ESES measures an individual's perceived ability to overcome various obstacles to perform physical activity.
Sleep Efficiency | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  Sleep efficiency is the total number of minutes of sleep divided by the number of minutes spent in bed. Sleep efficiency is measured by polysomnography.

SECONDARY OUTCOMES:
Functional Capacity | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  Functional capacity is evaluated using a Bruce protocol treadmill maximal exertion stress test. The maximum amount of work performed by the participant on the treadmill is measured as metabolic equivalents (METs)
Dynamic Gait Index (DGI) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A common clinical measure used to evaluate dynamic balance and coordination during a person's daily activities.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A self-reported measure to evaluate and monitor overall sleep quality.
Mayo Portland Adaptability Index (MPAI-4) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A measure of self-reported quality of life, limitation severity, and community participation after TBI.
Community Reintegration of Service Members (CRIS) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A self-reported measure of the ability of service members to reintegrate after returning to civilian life.

OTHER OUTCOMES:
California Verbal Learning Test-Second Edition (CVLT-II) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A widely used measure of verbal learning and memory using a multiple-trial list-learning task.
Brief Symptoms Inventory 18 (BSI-18) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A self-report measure of depression, anxiety, somatic concerns, and general distress.
Post-Traumatic Stress Disorder Checklist (PCL) | Change from baseline, after intervention (week 11), and 3 months after (week 24)
  A measure of the severity of PTSD related symptoms including intrusive thoughts, avoidance behavior, and arousal.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No